CLINICAL TRIAL: NCT05345964
Title: A Safety, Tolerability, Pharmacokinetics, and Food Impact Phase I Study of GST-HG151 Tablets in Single-dose and Multiple-dose in Healthy Volunteers
Brief Title: Phase I Study of GST-HG151 Tablets in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cosunter Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: GST-HG151-I-01
Record Dates: First submitted 2022-04-06; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single-dose experimental group (Active Comparator): 5mg,15mg,30mg,60mg,90mg,120mg,150mg and 180mg need to complete a single-dose clinical study. The first two dose groups had 4 subjects in each group (3 received GST-HG151 and 1 received placebo，randomly assigned), and the rest are 10 ubjects in each group (8 received GST-HG151 and 2 received placebo， randomly assigned)
  Interventions: Drug: GST-HG151
- Single-dose control group (Placebo Comparator): 5mg,15mg,30mg,60mg,90mg,120mg,150mg and 180mg need to complete a single-dose clinical study. The first two dose groups had 4 subjects in each group (3 received GST-HG151 and 1 received placebo，randomly assigned), and the rest are 10 ubjects in each group (8 received GST-HG151 and 2 received placebo， randomly assigned)
  Interventions: Drug: Placebo
- Multi-dose experimental group (Active Comparator): According to the results of the SAD, it is planned to carry out multiple-dose studies in 2 to 3 dose groups. Continuous administration, 12 subjects in each group(10 received GST-HG151 and 2 received placebo， randomly assigned)
  Interventions: Drug: GST-HG151
- Multi-dose control group (Placebo Comparator): According to the results of the SAD, it is planned to carry out multiple-dose studies in 2 to 3 dose groups. Continuous administration, 12 subjects in each group(10 received GST-HG151 and 2 received placebo， randomly assigned)
  Interventions: Drug: Placebo
- Food Impact Study Group A (Active Comparator): According to the results of the SAD, it is planned to select 1 dose group，10 subjects(8 received GST-HG151 and 2 received placebo， randomly assigned)，two cycles, crossover
  Interventions: Drug: GST-HG151
- Food Impact Study Group B (Active Comparator): According to the results of the SAD, it is planned to select 1 dose group，8 subjects，two cycles, crossover
  Interventions: Drug: GST-HG151

INTERVENTIONS:
Drug: GST-HG151 — Subjects will take GST-HG151 orally(once daily) on Day 1
  Arms: Single-dose experimental group
Drug: Placebo — Subjects will take Placebo orally(once daily) on Day 1
  Arms: Single-dose control group
Drug: GST-HG151 — Subjects will take GST-HG151 orally (once daily) from Day 1 to Day 7
  Arms: Multi-dose experimental group
Drug: Placebo — Subjects will take Placebo orally (once daily) from day 1 to day 7
  Arms: Multi-dose control group
Drug: GST-HG151 — Group A was administered under the fasting condition of Day1 in the first cycle, and under the postprandial conditions of Day8 ~ Day15 in the second cycle. The two cycles are cross-administered, and the cleaning period is 7 to 14 days.
  Arms: Food Impact Study Group A
Drug: GST-HG151 — Group B was administered under the postprandial conditions of Day1 in the first cycle, and under the sky-abdominal conditions of Day8 ~ Day15 in the second cycle. The two cycles are cross-administered, and the cleaning period is 7 to 14 days.
  Arms: Food Impact Study Group B

SUMMARY:
To Evaluate the Safety, Tolerability, Pharmacokinetics, and Food Impact of GST-HG151 Tablets in Single-dose and Multiple-dose in Healthy Volunteers

DETAILED DESCRIPTION:
This trial includes single-dose studies,multiple-dose studies and food Impact studies, The single-dose study included eight doses groups of 5 mg, 15 mg, 30 mg, 60 mg, 90mg, 120 mg, 150 mg and 180 mg. Based on the results of a single dose, select 2 to 3 doses to conduct multiple dose studies. To evaluate the tolerance of GST-HG131 tablets in healthy subjects in single and multiple administrations, pharmacokinetic characteristics, drug metabolism and transformation, and the effect of food on GST-HG151 pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial and fully understand the content, process and possible adverse reactions of the trial.
2. Subjects (including partners) are willing to take effective pregnancy avoidance measures within 6 months after screening to the last study drug administration.
3. Male and female healthy subjects aged 18 to 45 years (including 18 and 45 years old).
4. Male subjects weigh no less than 50 kg, and female subjects weigh no less than 45 kg. Body mass index (BMI) = body weight (kg) / height 2 (m2), body mass index is in the range of 19 ~ 24 kg / m2 (including critical value).
5. Good physical condition (no significant clinical symptoms, normal physical examination. no clinically significant of laboratory examination, vital signs, 12 lead ECG, chest film and abdominal B-ultrasound results).

Exclusion Criteria:

1. Allergic constitution (allergic to a variety of drugs, especially ingredients similar to the test drug, or excipients of the test drug, or food).
2. Smokers or those who smoke more than 5 cigarettes per day in the three months before screening, or disagree to avoid using any tobacco products during the study.
3. Have a history of alcoholism or drink regularly in the three months before screening, those who drink more than 14 units of alcohol per week (1 unit = 360ml of beer with 5% alcohol content or 45ml of spirits with 40% alcohol content or 150ml of wine with 12% alcohol content). Who cannot stop alcohol intake during the study or have a positive breath test for alcoho.
4. Blood donation or massive blood loss (≥300 mL, , except female menstruation) or use blood products or blood transfusion within 3 months before screening.
5. Have special requirements for diet and cannot abide by the unified diet.
6. Took any prescription drugs, over-the-counter drugs, health products or Chinese herbal medicine within 2 weeks before screening.
7. Have taken the study drug or participated in the drug clinical trial within three months before taking the study drug(Except for those who did not enter the group).
8. Take any drugs that alter liver enzyme activity CYP3A4, including strong inhibitors and inducers that affect CYP3A4, within 28 days before screening or during the study.
9. Female subjects were breastfeeding during the screening period or during the trial or were preparing for pregnancy recently or had a positive serum pregnancy result.
10. Have been smoking,drinking,or Ingested tea, any caffeinated or xanthine-rich food or drink,or special diet (including dragon fruit, mango, grapefruit, etc.),or have vigorous exercise, or have other factors affecting drug absorption, distribution, metabolism, excretion, etc.within 48hours before screening.
11. Ingested chocolate,any alcohol-containing product within 24 hours before screening.
12. Subjects who cannot tolerate the standard meal (high fat and high calorie meal) (this strip is only applicable to subjects participating in the food impact study).
13. Have a history of dysphagia or any gastrointestinal disease that affects drug absorption.
14. Clinical laboratory examinations are abnormal and clinically significant, or the following diseases (including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, Immune, mental or cardiovascular disease).
15. HBsAg, HCV, HIV and TPPA have one or more positive.
16. had undergone major surgery within 4 weeks before screening or planned surgery during the trial.
17. Have a history of drug abuse, or have used drugs within 3 months before screening, or those who are positive in the screening test of urine drugs and drugs (methamphetamine, tetrahydrocannabinol acid, ketamine, cocaine, benzodiazepine, dimethylbisoxyamphetamine and morphine).
18. Have difficulty in blood collection, or have a history of needle fainting or cannot tolerate venipuncture.
19. Cannot complete the trial for other reasons, or the investigator believes should not be included.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
AEs and SAEs | SAD Cohorts : Up to Day 6. MAD Cohorts : Up to Day 14. Food Effect Cohorts : Up to Day 20.
  Safety assessments such as AEs and SAEs
Peak Plasma Concentration (Cmax) | Before and at pre-specified time points up to 72 hours after dosing.
  Plasma samples were collected at different points for pharmacokinetic analysis
Area Under Curve (AUC) | Before and at pre-specified time points up to 72 hours after dosing.
  Plasma samples were collected at different points for pharmacokinetic analysis
T1/2 | Before and at pre-specified time points up to 72 hours after dosing.
  Plasma samples were collected at different points for pharmacokinetic analysis
Cl/F | Before and at pre-specified time points up to 72 hours after dosing.
  Plasma samples were collected at different points for pharmacokinetic analysis
Ae | Before and at pre-specified time points up to 72 hours after dosing.
  Plasma samples were collected at different points for pharmacokinetic analysis
Fe | Before and at pre-specified time points up to 72 hours after dosing.
  Plasma samples were collected at different points for pharmacokinetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ling Zheng, Bachelor, Principal Investigator — Mengchao Hepatpbiliary Hospital of Fujian Medical University
Locations (1):
- Mengchao Hepatpbiliary Hospital of Fujian Medical University, Fujian, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No